CLINICAL TRIAL: NCT05048394
Title: Teleoperation Experimental Comparison With Able-bodied Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Point Designs (Industry)
Collaborators: University of Colorado, Boulder (Other); National Institute for Biomedical Imaging and Bioengineering (NIBIB) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Device Feasibility
Other Study IDs: 377394; R41EB032723 (NIH)
Record Dates: First submitted 2021-09-08; First posted 2021-09-17 (Actual); Results first posted 2024-12-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Amputation; Traumatic, Arm, Upper

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Standard-of-care then Semi-autonomous myoelectric control (Experimental): The standard of care myoelectric control algorithm will be implemented on a by-pass prosthetic socket with a sensorized TASKA prosthetic hand
  The semi-autonomous myoelectric control algorithm will be implemented on a by-pass prosthetic socket with a sensorized TASKA prosthetic hand.
  Interventions: Device: Semi-autonomous myoelectric control algorithm; Device: Standard-of-care myoelectric control algorithm
- Semi-autonomous then Standard-of-care myoelectric control (Experimental): The semi-autonomous myoelectric control algorithm will be implemented on a by-pass prosthetic socket with a sensorized TASKA prosthetic hand.
  The standard of care myoelectric control algorithm will be implemented on a by-pass prosthetic socket with a sensorized TASKA prosthetic hand
  Interventions: Device: Semi-autonomous myoelectric control algorithm; Device: Standard-of-care myoelectric control algorithm

INTERVENTIONS:
Device: Semi-autonomous myoelectric control algorithm — The semi-autonomous myoelectric control algorithm will be implemented on a by-pass prosthetic socket with a sensorized TASKA prosthetic hand.
Device: Standard-of-care myoelectric control algorithm — The standard of care myoelectric control algorithm will be implemented on a by-pass prosthetic socket with a sensorized TASKA prosthetic hand.

SUMMARY:
To compare the use of the semi-autonomous control algorithm (condition 1) with the standard of care myoelectric system used with the TASKA prosthetic hand (condition 2). Able bodied subjects will enroll in a laboratory based experimental session at the University of Colorado at Boulder. Subjects will be fitted with a by-pass prosthesis which enables the able-bodied subject to control the prosthetic hand using the myoelectric signals on their able limb. A TASKA prosthetic hand will be sensorized using the Point Touch technology. In a randomized order, the subjects will perform functional tasks evaluating dexterity and assistance with prolonged gross motor movement using each experimental condition. Then, a direct comparison can be made across subjects for the semi-autonomous control algorithm and the standard of care myoelectric system used in the TASKA prosthetic hand.

ELIGIBILITY:
Inclusion Criteria:

* Able-bodied subject
* Fluent in English
* Age of 18 years or greater

Exclusion Criteria:

* Significant cognitive deficits as determined upon clinical evaluation
* Significant neurological deficits as determined upon clinical evaluation
* Significant physical deficits of the residual limb impacting full participation in the study as determined upon clinical evaluation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Colorado Boulder, Boulder, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard-of-care Then Semi-autonomous Myoelectric Control: The standard of care myoelectric control algorithm will be implemented on a by-pass prosthetic socket with a sensorized TASKA prosthetic hand
  The semi-autonomous myoelectric control algorithm will be implemented on a by-pass prosthetic socket with a sensorized TASKA prosthetic hand.
  Semi-autonomous myoelectric control algorithm: The semi-autonomous myoelectric control algorithm will be implemented on a by-pass prosthetic socket with a sensorized TASKA prosthetic hand.
  Standard-of-care myoelectric control algorithm: The standard of care myoelectric control algorithm will be implemented on a by-pass prosthetic socket with a sensorized TASKA prosthetic hand.
- Semi-autonomous Then Standard-of-care Myoelectric Control: The semi-autonomous myoelectric control algorithm will be implemented on a by-pass prosthetic socket with a sensorized TASKA prosthetic hand.
  The standard of care myoelectric control algorithm will be implemented on a by-pass prosthetic socket with a sensorized TASKA prosthetic hand
  Semi-autonomous myoelectric control algorithm: The semi-autonomous myoelectric control algorithm will be implemented on a by-pass prosthetic socket with a sensorized TASKA prosthetic hand.
  Standard-of-care myoelectric control algorithm: The standard of care myoelectric control algorithm will be implemented on a by-pass prosthetic socket with a sensorized TASKA prosthetic hand.
Period: Overall Study
Arm/Group | Standard-of-care Then Semi-autonomous Myoelectric Control | Semi-autonomous Then Standard-of-care Myoelectric Control
Started | 7 | 4
Completed | 7 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard-of-care Then Semi-autonomous Myoelectric Control | Semi-autonomous Then Standard-of-care Myoelectric Control | Total
Number analyzed (Participants) | 7 | 4 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 4 | 11
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 30 (7) | 27 (1) | 29 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 5 | 3 | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 7 | 4 | 14
Handedness [Count of Participants; unit: Participants] — Dominant hand of participants
  Participants
    Right | 6 | 3 | 9
    Left | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Transfer Success Rate in a Fragile Box and Blocks Task
Description: The participant is instructed to transfer a fragile, ball-like object that breaks at 8 Newtons of force over a 10-centimeter high barrier as many times as possible in a 2-minute period. A broken or dropped object is considered an unsuccessful transfer. The number of successful and attempted transfers is recorded. This task is modeled after the Box-and-Blocks Test and has been used to validate fine dexterity of myoelectric upper limb prostheses.
Time Frame: Day 1 (1 hour)
Measure: Mean (Standard Deviation); unit: percentage of attempted transfers
Arm/Group | Standard-of-care Then Semi-autonomous Myoelectric Control | Semi-autonomous Then Standard-of-care Myoelectric Control
Number analyzed (Participants) | 7 | 4
percentage of attempted transfers
  Standard-of-care control | 67.50 (20.35) | 72.75 (17.54)
  Semi-autonomous control | 93.46 (9.02) | 95.06 (6.93)
Statistical Analysis 1: Comparison: Standard-of-care Then Semi-autonomous Myoelectric Control vs Semi-autonomous Then Standard-of-care Myoelectric Control; Test type: Equivalence — Equivalence is defined as a difference of 0; p < 0.001, Wilcoxon (Mann-Whitney) — Threshold for statistical significance was p = 0.05

2. Secondary Outcome: Ball Drops in a Holding Task
Description: The participant is instructed to pick up a 2-inch Styrofoam ball and hold the object above the desk or table for 2 minutes. If the ball is dropped, the participant is instructed to pick it back up. The 2-minute timer does not restart. The number of times the ball was dropped is recorded. This task has been used to validate the ability of myoelectric prostheses to assist with gross, prolonged movements.
Time Frame: Day 1 (1 hour)
Measure: Median (Full Range); unit: ball drops
Arm/Group | Standard-of-care Then Semi-autonomous Myoelectric Control | Semi-autonomous Then Standard-of-care Myoelectric Control
Number analyzed (Participants) | 7 | 4
ball drops
  Standard-of-care control | 0 [0 to 1] | 0 [0 to 1]
  Semi-autonomous control | 1 [0 to 2] | 0 [0 to 2]
Statistical Analysis 1: Comparison: Standard-of-care Then Semi-autonomous Myoelectric Control vs Semi-autonomous Then Standard-of-care Myoelectric Control; Test type: Equivalence — Equivalence is defined as a difference of 0; p = 0.14, Wilcoxon (Mann-Whitney) — Threshold for significance was p = 0.05

ADVERSE EVENTS:
Time Frame: 9 days
Arm/Group | Standard-of-care Then Semi-autonomous Myoelectric Control | Semi-autonomous Then Standard-of-care Myoelectric Control
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/4
Other Adverse Events (participants affected / at risk) | 0/7 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-07-19): https://cdn.clinicaltrials.gov/large-docs/94/NCT05048394/Prot_000.pdf
  • Statistical Analysis Plan (2024-11-27): https://cdn.clinicaltrials.gov/large-docs/94/NCT05048394/SAP_001.pdf